CLINICAL TRIAL: NCT06779968
Title: Multimodal Analgesia Versus Peripheral Nerve Block for Postoperative Pain Management After Lower Limb Injury Surgery: a Randomized Controlled Trial
Brief Title: Multimodal Analgesia Versus Peripheral Nerve Block for Postoperative Pain Management After Lower Limb Injury Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaguang Duan (Other)
Responsible Party: Sponsor-Investigator, Xiaguang Duan, Deputy Chief of Anesthesiology, Inner Mongolia Baogang Hospital
Organization: Inner Mongolia Baogang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-MER-317
Record Dates: First submitted 2025-01-14; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Lower Limb Injury
MeSH Terms: conditions — Leg Injuries | interventions — Analgesia, Epidural; Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (5):
- FNB Group (Experimental): In the femoral nerve block (FNB) group, the femoral nerve was blocked distal to the inguinal ligament and lateral to the femoral artery. Under sterile conditions and ultrasound guidance using a short-axis out-of-plane approach, a 22-gauge insulated needle was advanced adjacent to the femoral nerve. Following confirmation of correct needle tip placement, a 20 mL volume of either 266 mg liposomal bupivacaine (diluted as indicated) or 0.2% ropivacaine was injected. This was followed by a continuous infusion at a rate of 5-10 mL/hr. For pediatric patients, a continuous infusion of 0.2% ropivacaine was administered at an initial bolus of 0.2-0.5 mg/kg, followed by a continuous infusion of 0.1-0.3 mg/kg/hr.
  Interventions: Device: Femoral Nerve Block; Device: General Aneasthesia
- CS-FNB Group (Experimental): In the combined sciatic and femoral nerve block (CS-FNB) group, the femoral nerve block was performed as described above. The sciatic nerve block was performed at either the gluteal region or popliteal fossa. Under sterile conditions and ultrasound guidance using either an in-plane or out-of-plane approach, a 22-gauge insulated needle was advanced adjacent to the sciatic nerve. Following confirmation of correct needle tip placement, a 20 mL volume of either 266 mg liposomal bupivacaine (diluted as indicated) or 0.2% ropivacaine was injected. This was followed by a continuous infusion at a rate of 5-10 mL/hr. For pediatric patients, a continuous infusion of 0.2% ropivacaine was administered at an initial bolus of 0.2-0.5 mg/kg, followed by a continuous infusion of 0.1-0.3 mg/kg/hr.
  Interventions: Device: Combined Sciatic and Femoral Nerve Block; Device: General Aneasthesia
- LPB Group (Experimental): In the lumbar plexus block (LPB) group, the lumbar plexus was blocked paraspinally within the psoas muscle. Under sterile conditions, ultrasound guidance, or with the assistance of a nerve stimulator, using either an in-plane or out-of-plane approach, a 22-gauge insulated needle was advanced within the psoas muscle adjacent to the lumbar plexus. Following confirmation of correct needle tip placement, a 20 mL volume of either 266 mg liposomal bupivacaine (diluted as indicated) or 0.2% ropivacaine was injected. This was followed by a continuous infusion at a rate of 5-10 mL/hr. For pediatric patients, a continuous infusion of 0.2% ropivacaine was administered at an initial bolus of 0.2-0.5 mg/kg, followed by a continuous infusion of 0.1-0.3 mg/kg/hr.
  Interventions: Device: Lumbar plexus block; Device: General Aneasthesia
- EA group (Active Comparator): For epidural analgesia, an initial bolus of 5-15 mL of 0.5% ropivacaine was administered followed by a continuous infusion of 0.2% ropivacaine at a rate of 3-10 mL/hr. For pediatric patients, an initial bolus of 0.2% ropivacaine at 0.5-1 mg/kg was administered, not exceeding a maximum total dose of 2-2.5 mg/kg, followed by a continuous infusion of 0.1-0.3 mg/kg/hr.
  Interventions: Procedure: Epidural Analgesia
- PCA group (Experimental): For intravenous patient-controlled analgesia (PCA), fentanyl was administered at a dose of 2 mcg/kg, diluted in 100 mL of normal saline. The basal infusion rate was set at 2 mL/hr, with a PCA dose of 2 mL and a lockout interval of 15 minutes.
  Interventions: Drug: Intravenous patient-controlled analgesia; Device: General Aneasthesia

INTERVENTIONS:
Device: Femoral Nerve Block — In the femoral nerve block (FNB) group, the femoral nerve was blocked distal to the inguinal ligament and lateral to the femoral artery. Under sterile conditions and ultrasound guidance using a short-axis out-of-plane approach, a 22-gauge insulated needle was advanced adjacent to the femoral nerve. Following confirmation of correct needle tip placement, a 20 mL volume of either 266 mg liposomal bupivacaine (diluted as indicated) or 0.2% ropivacaine was injected. This was followed by a continuous infusion at a rate of 5-10 mL/hr. For pediatric patients, a continuous infusion of 0.2% ropivacaine was administered at an initial bolus of 0.2-0.5 mg/kg, followed by a continuous infusion of 0.1-0.3 mg/kg/hr.
  Arms: FNB Group
Device: Combined Sciatic and Femoral Nerve Block — In the combined sciatic and femoral nerve block (CS-FNB) group, the femoral nerve block was performed as described above. The sciatic nerve block was performed at either the gluteal region or popliteal fossa. Under sterile conditions and ultrasound guidance using either an in-plane or out-of-plane approach, a 22-gauge insulated needle was advanced adjacent to the sciatic nerve. Following confirmation of correct needle tip placement, a 20 mL volume of either 266 mg liposomal bupivacaine (diluted as indicated) or 0.2% ropivacaine was injected. This was followed by a continuous infusion at a rate of 5-10 mL/hr. For pediatric patients, a continuous infusion of 0.2% ropivacaine was administered at an initial bolus of 0.2-0.5 mg/kg, followed by a continuous infusion of 0.1-0.3 mg/kg/hr.
  Arms: CS-FNB Group
Device: Lumbar plexus block — In the lumbar plexus block (LPB) group, the lumbar plexus was blocked paraspinally within the psoas muscle. Under sterile conditions, ultrasound guidance, or with the assistance of a nerve stimulator, using either an in-plane or out-of-plane approach, a 22-gauge insulated needle was advanced within the psoas muscle adjacent to the lumbar plexus. Following confirmation of correct needle tip placement, a 20 mL volume of either 266 mg liposomal bupivacaine (diluted as indicated) or 0.2% ropivacaine was injected. This was followed by a continuous infusion at a rate of 5-10 mL/hr. For pediatric patients, a continuous infusion of 0.2% ropivacaine was administered at an initial bolus of 0.2-0.5 mg/kg, followed by a continuous infusion of 0.1-0.3 mg/kg/hr.
  Arms: LPB Group
Procedure: Epidural Analgesia — For epidural analgesia, an initial bolus of 5-15 mL of 0.5% ropivacaine was administered followed by a continuous infusion of 0.2% ropivacaine at a rate of 3-10 mL/hr. For pediatric patients, an initial bolus of 0.2% ropivacaine at 0.5-1 mg/kg was administered, not exceeding a maximum total dose of 2-2.5 mg/kg, followed by a continuous infusion of 0.1-0.3 mg/kg/hr.
  Arms: EA group
Drug: Intravenous patient-controlled analgesia — For intravenous patient-controlled analgesia (PCA), fentanyl was administered at a dose of 2 mcg/kg, diluted in 100 mL of normal saline. The basal infusion rate was set at 2 mL/hr, with a PCA dose of 2 mL and a lockout interval of 15 minutes.
  Arms: PCA group
Device: General Aneasthesia — Following administration of the regional anesthesia, general anesthesia with endotracheal intubation will be performed. Anesthesia induction will be achieved using propofol (1.5-2 mg/kg i.v.), rocuronium (1-2 mg/kg i.v.), and fentanyl (1-2 μg/kg i.v.). Anesthesia will be maintained using sevoflurane or desflurane, with inhaled concentration adjusted based on Bispectral Index (BIS) monitoring. A continuous infusion of remifentanil (0.05-0.2 μg/kg/min) will be administered, with adjustments to maintain blood pressure and heart rate within ±20% of baseline values. Following induction, patients will be mechanically ventilated in pressure-regulated volume control (PRVC) mode. The ventilator (Aestiva; GE Healthcare, Waukesha, Wisconsin, USA) settings will be: tidal volume 6-8 mL/kg, positive end-expiratory pressure 0 cm H2O, inspiratory to expiratory ratio 1:2, respiratory rate 16 breaths per minute (BPM), and fraction of inspired oxygen 41%.
  Arms: CS-FNB Group; FNB Group; LPB Group; PCA group

SUMMARY:
The purpose of this clinical trial is to understand the effectiveness of femoral nerve block, combined sciatic and femoral nerve block, lumbar plexus block, epidural block, and intravenous analgesia pump in the application of lower limb injury (total knee replacement, knee arthroscopy, patella fracture, femoral shaft fracture) surgery. It will also understand the safety of the drugs liposomal bupivacaine and ropivacaine. The main question it aims to answer is: Does nerve block reduce the number of times participants need to use analgesics postoperatively? The researchers will compare femoral nerve block, combined sciatic and femoral nerve block, lumbar plexus block, epidural block, and intravenous analgesia pump to see which analgesic method has the best postoperative analgesic effect. Participants will: undergo nerve block first, then endotracheal intubation general anesthesia after entering the operating room; record vital signs during surgery, record postoperative analgesic doses, NRS pain scores, patient satisfaction, and postoperative nausea and vomiting.

DETAILED DESCRIPTION:
Study Design: This study was a prospective, randomized, controlled, comparative clinical trial with both participant and clinician blinding. This trial was designed to assess both the superiority and non-inferiority of different analgesic modalities in the management of postoperative pain following lower limb surgery. The study evaluated the effectiveness of femoral nerve block, combined sciatic and femoral nerve block, lumbar plexus block, epidural analgesia, and intravenous patient-controlled analgesia for patients undergoing procedures such as total knee replacement, knee arthroscopy, patella fracture repair, and pediatric femoral shaft fracture repair. Participants were recruited from Baogang Hospital, Inner Mongolia. This study received approval from the Medical Ethics Committee of Baogang Hospital, Inner Mongolia, and was conducted in accordance with the principles of the Declaration of Helsinki and the Consolidated Standards of Reporting Trials (CONSORT) guidelines. All participants provided informed written consent.

Patients：A total of 150 patients, classified as American Society of Anesthesiologists (ASA) physical status I, II, or III and aged 2 years or older, undergoing postoperative analgesia for lower limb injuries were recruited between February 2025 and May 2025. Participants were randomly assigned to one of five study groups, with 30 participants in each group.

Randomization and Blinding：This study employed block randomization to generate the random allocation sequence. A block size of 6 was set, and the random sequence was generated using dedicated software (the blockrand package in R version 4.3.2). The allocation of the random sequence was performed by an independent third party, and allocation concealment was implemented using sequentially numbered, sealed, opaque envelopes. The research team remained blinded throughout the randomization process and was not involved in the generation or allocation of the random sequence.

Intervention： Upon arrival to the operating room, patients will be monitored with electrocardiography, blood pressure, and pulse oximetry. Patients will be placed in the prone position with their arms abducted and internally rotated. Ultrasound guidance will be used for all regional anesthesia procedures (SonoSite Edge II; Fujifilm SonoSite, Bothell, WA, USA) with a linear 13-6 MHz ultrasound probe (HFL50x; Fujifilm SonoSite, Bothell, WA, USA). For each block, a 5 mL test dose will be injected initially, followed by observation for clinical signs of a successful block. After confirming correct placement, the remaining dose of the anesthetic agent will be injected. Following administration of the regional anesthesia, general anesthesia with endotracheal intubation will be performed. Anesthesia induction will be achieved using propofol (1.5-2 mg/kg i.v.), rocuronium (1-2 mg/kg i.v.), and fentanyl (1-2 μg/kg i.v.). Anesthesia will be maintained using sevoflurane or desflurane, with inhaled concentration adjusted based on Bispectral Index (BIS) monitoring. A continuous infusion of remifentanil (0.05-0.2 μg/kg/min) will be administered, with adjustments to maintain blood pressure and heart rate within ±20% of baseline values. Following induction, patients will be mechanically ventilated in pressure-regulated volume control (PRVC) mode. The ventilator (Aestiva; GE Healthcare, Waukesha, Wisconsin, USA) settings will be: tidal volume 6-8 mL/kg, positive end-expiratory pressure 0 cm H2O, inspiratory to expiratory ratio 1:2, respiratory rate 16 breaths per minute (BPM), and fraction of inspired oxygen 41%.

Femoral Nerve Block (FNB) Group: In the femoral nerve block (FNB) group, the femoral nerve was blocked distal to the inguinal ligament and lateral to the femoral artery. Under sterile conditions and ultrasound guidance using a short-axis out-of-plane approach, a 22-gauge insulated needle was advanced adjacent to the femoral nerve. Following confirmation of correct needle tip placement, a 20 mL volume of either 266 mg liposomal bupivacaine (diluted as indicated) or 0.2% ropivacaine was injected. This was followed by a continuous infusion at a rate of 5-10 mL/hr. For pediatric patients, a continuous infusion of 0.2% ropivacaine was administered at an initial bolus of 0.2-0.5 mg/kg, followed by a continuous infusion of 0.1-0.3 mg/kg/hr.

Combined Sciatic and Femoral Nerve Block (CS-FNB) Group: In the combined sciatic and femoral nerve block (CS-FNB) group, the femoral nerve block was performed as described above. The sciatic nerve block was performed at either the gluteal region or popliteal fossa. Under sterile conditions and ultrasound guidance using either an in-plane or out-of-plane approach, a 22-gauge insulated needle was advanced adjacent to the sciatic nerve. Following confirmation of correct needle tip placement, a 20 mL volume of either 266 mg liposomal bupivacaine (diluted as indicated) or 0.2% ropivacaine was injected. This was followed by a continuous infusion at a rate of 5-10 mL/hr. For pediatric patients, a continuous infusion of 0.2% ropivacaine was administered at an initial bolus of 0.2-0.5 mg/kg, followed by a continuous infusion of 0.1-0.3 mg/kg/hr.

Lumbar Plexus Block (LPB) Group: In the lumbar plexus block (LPB) group, the lumbar plexus was blocked paraspinally within the psoas muscle. Under sterile conditions, ultrasound guidance, or with the assistance of a nerve stimulator, using either an in-plane or out-of-plane approach, a 22-gauge insulated needle was advanced within the psoas muscle adjacent to the lumbar plexus. Following confirmation of correct needle tip placement, a 20 mL volume of either 266 mg liposomal bupivacaine (diluted as indicated) or 0.2% ropivacaine was injected. This was followed by a continuous infusion at a rate of 5-10 mL/hr. For pediatric patients, a continuous infusion of 0.2% ropivacaine was administered at an initial bolus of 0.2-0.5 mg/kg, followed by a continuous infusion of 0.1-0.3 mg/kg/hr.

Epidural Analgesia: For epidural analgesia, an initial bolus of 5-15 mL of 0.5% ropivacaine was administered followed by a continuous infusion of 0.2% ropivacaine at a rate of 3-10 mL/hr. For pediatric patients, an initial bolus of 0.2% ropivacaine at 0.5-1 mg/kg was administered, not exceeding a maximum total dose of 2-2.5 mg/kg, followed by a continuous infusion of 0.1-0.3 mg/kg/hr.

Intravenous Patient-Controlled Analgesia (PCA): For intravenous patient-controlled analgesia (PCA), fentanyl was administered at a dose of 2 mcg/kg, diluted in 100 mL of normal saline. The basal infusion rate was set at 2 mL/hr, with a PCA dose of 2 mL and a lockout interval of 15 minutes.

Outcomes and measures：Participants were followed up in the ward by two specially trained research nurses who were blinded to the participants' treatment group assignments. Outcome assessments were conducted at the following time points: prior to treatment (baseline), 2 hours postoperatively, 6 hours postoperatively, 12 hours postoperatively, and 24 hours postoperatively. These assessments were performed either in person or via telephone.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status classification I-III
* Patients (or their guardians) voluntarily participate in this study and sign a written informed consent form
* Patients (or their guardians) are able to understand the study content and cooperate with the study protocol

Exclusion Criteria:

* Known allergy to local anesthetics or opioid analgesics.
* Presence of contraindications to local or epidural anesthesia.
* Presence of undiagnosed or poorly characterized neuropathic pain.
* Presence of severe mental illness that would impede the participant's ability to cooperate with study assessment and treatment procedures.
* Clinically significant coagulopathy or current use of anticoagulant medications.
* Presence of infection at the planned puncture site or systemic infection.
* Pregnancy or lactation.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale(NRS) | At baseline (before therapy), at 2 hours post-treatment, at 6 hours post-treatment, at 12 hours post-treatment, and at 24 hours post-treatment
  The NRS, Numerical Rating Scale, is a rating system from 0 to 10, where 0 represents "no pain" and 10 represents the worst possible pain.

SECONDARY OUTCOMES:
Postoperative Opioid Consumption | Total consumption measured at 24 hours post-treatment and at 48 hours post-treatment.
  This measure records the total amount of opioid medication (e.g., fentanyl) consumed by the patient post-operatively. Both intravenous (via PCA) and oral opioid consumption will be recorded in total.
Postoperative Nausea and Vomiting (PONV) | At 2 hours post-treatment, at 6 hours post-treatment, at 12 hours post-treatment and at 24 hours post-treatment.
  PONV is assessed by recording the presence or absence of nausea and vomiting. If present, the severity of nausea will be evaluated using a qualitative scale (e.g., none, mild, moderate, severe) or a scoring system such as the PONV score. The occurrence of vomiting will be recorded as a binary (yes/no) variable.
Patient Satisfaction | At 48 hours post-treatment.
  Patient satisfaction with the pain management method is assessed using a standardized questionnaire, which includes questions about their perceived level of pain control, comfort with the analgesic technique, and their willingness to choose the same method again in the future, measured by a likert scale score (e.g. 1=Strongly Disagree, 5=Strongly Agree).

CONTACTS AND LOCATIONS:
Locations (1):
- Inner Mongolia Baogang Hospital, Baotou, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: January 2026-January 2031
Access Criteria: A proposal that describes planned analyses must be submitted or whether a data sharing agreement must be signed.